CLINICAL TRIAL: NCT06446388
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of QLS31905 and/or QL1706 Combination Chemotherapy for the Treatment of CLDN18.2-Positive Advanced Malignant Solid Tumors
Brief Title: Study of QLS31905 and/or QL1706 Combination With Chemotherapy in the Advanced Malignant Solid Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLS31905-202
Record Dates: First submitted 2024-06-01; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Oxaliplatin; Capecitabine; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- QLS31905 + oxaliplatin + capecitabine (Experimental): Gastric/gastroesophageal junction cancer participants will be treated with QLS31905 at doses determined by the phase I study in combination with oxaliplatin and capecitabine.
  Interventions: Drug: QLS31905; Drug: Oxaliplatin; Drug: Capecitabine
- QL1706 + oxaliplatin + capecitabine (Experimental): Gastric/gastroesophageal junction cancer participants will be treated with QL1706 in combination with oxaliplatin and capecitabine.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: QL1706
- QLS31905 + oxaliplatin + capecitabine + QL1706 (Experimental): Gastric/gastroesophageal junction cancer participants will be treated with QLS31905 at doses determined by the phase I study in combination with oxaliplatin and capecitabine+ QL1706.
  Interventions: Drug: QLS31905; Drug: Oxaliplatin; Drug: Capecitabine; Drug: QL1706
- QLS31905 + gemcitabine+cisplatin (Experimental): Biliary tract cancer will be treated with QLS31905 at doses determined by the phase I study in combination with gemcitabine and cisplatin.
  Interventions: Drug: QLS31905; Drug: Gemcitabine; Drug: Cisplatin
- QL1706 + gemcitabine+cisplatin (Experimental): Biliary tract cancer will be treated with QL1706 in combination with gemcitabine and cisplatin.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: QL1706
- QLS31905 + gemcitabine+cisplatin+ QL1706 (Experimental): Biliary tract cancer will be treated with QLS31905 at doses determined by the phase I study in combination with gemcitabine and cisplatin+ QL1706.
  Interventions: Drug: QLS31905; Drug: Gemcitabine; Drug: Cisplatin; Drug: QL1706
- QLS31905 + standard chemotherapy (Experimental): Other solid tumor participants will be treated with QLS31905 at doses determined by the phase I study in combination with standard chemotherapy recommended by guidelines.
  Interventions: Drug: QLS31905; Drug: Chemotherapy drug
- QL1706 + standard chemotherapy (Experimental): Other solid tumor participants will be treated with QL1706 in combination with standard chemotherapy recommended by guidelines.
  Interventions: Drug: QL1706; Drug: Chemotherapy drug
- QLS31905 + standard chemotherapy + QL1706 (Experimental): Other solid tumor participants will be treated with QLS31905 at doses determined by the phase I study in combination with standard chemotherapy and QL1706.
  Interventions: Drug: QLS31905; Drug: QL1706; Drug: Chemotherapy drug

INTERVENTIONS:
Drug: QLS31905 — Administered as an intravenous infusion.
  Arms: QLS31905 + gemcitabine+cisplatin; QLS31905 + gemcitabine+cisplatin+ QL1706; QLS31905 + oxaliplatin + capecitabine; QLS31905 + oxaliplatin + capecitabine + QL1706; QLS31905 + standard chemotherapy; QLS31905 + standard chemotherapy + QL1706
Drug: Oxaliplatin — 130 mg/m2, intravenous infusion, D1, up to 8 cycles.
  Arms: QL1706 + oxaliplatin + capecitabine; QLS31905 + oxaliplatin + capecitabine; QLS31905 + oxaliplatin + capecitabine + QL1706
Drug: Capecitabine — 1000 mg/m2, oral, bid, D1-D14
  Arms: QL1706 + oxaliplatin + capecitabine; QLS31905 + oxaliplatin + capecitabine; QLS31905 + oxaliplatin + capecitabine + QL1706
Drug: Gemcitabine — 1000 mg/m2 administered as IV infusion on D1/D8 of each cycle.
  Arms: QL1706 + gemcitabine+cisplatin; QLS31905 + gemcitabine+cisplatin; QLS31905 + gemcitabine+cisplatin+ QL1706
Drug: Cisplatin — 25 mg/m2, intravenous infusion, D1/D8, up to 8 cycles.
  Arms: QL1706 + gemcitabine+cisplatin; QLS31905 + gemcitabine+cisplatin; QLS31905 + gemcitabine+cisplatin+ QL1706
Drug: QL1706 — 5 mg/kg, intravenous infusion,D1
  Arms: QL1706 + gemcitabine+cisplatin; QL1706 + oxaliplatin + capecitabine; QL1706 + standard chemotherapy; QLS31905 + gemcitabine+cisplatin+ QL1706; QLS31905 + oxaliplatin + capecitabine + QL1706; QLS31905 + standard chemotherapy + QL1706
Drug: Chemotherapy drug — Standard chemotherapy recommended by guidelines.
  Arms: QL1706 + standard chemotherapy; QLS31905 + standard chemotherapy; QLS31905 + standard chemotherapy + QL1706

SUMMARY:
This study aims to evaluate the efficacy and safety of QLS31905 and/or QL1706 plus chemotherapy in patients with Claudin18.2-positive advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in the study and sign the informed consent form;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1;
* Expected survival time ≥ 3 months;
* Histologically or cytologically confirmed locally advanced unresectable or metastatic solid tumors;
* No prior systemic anti-tumor treatment for locally advanced unresectable or metastatic disease;
* Tumor tissue samples determined to be positive for Claudin18.2 by immunohistochemistry (IHC);
* At least one measurable lesion per RECIST v1.1;
* Patients with adequate cardiac, liver, renal function, etc.

Exclusion Criteria:

* History of malignancies other than the target cancer within 5 years prior to the first dose of the investigational product ;
* Underwent major organ surgery (excluding needle biopsy) or had significant trauma within 28 days prior to enrollment, or requires elective surgery during the study;
* Known central nervous system metastases;
* Patients with hepatitis B; patients with hepatitis C; patients who test positive for syphilis, or patients with a known history of HIV or positive HIV screening test; Patients with a known history of psychoactive drug abuse, alcohol abuse, or substance abuse;
* Patients with added risks associated with the study or may interfere with the interpretation of study results as determined by the investigator, or deemed unsuitable by the investigator and/or sponsor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Approximately 24 months
  ORR is defined as the proportion of participants who have a best overall response of Complete Response (CR) or Partial Response (PR)

SECONDARY OUTCOMES:
Safety assessed by Adverse Events (AEs) | Approximately 24 months
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom,or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Safety assessed by incidence of serious adverse events (SAE) | Approximately 24 months
  Adverse Event (AE) is considered "serious" if the investigator or sponsor view any of the following outcomes: Death, life-threatening, persistent or significant disability/incapacity, congenital anomaly or birth defect,hospitalization, or medically important event.
Number of participants with laboratory value abnormalities | Approximately 24 months
  Number of participants with potentially clinically significant laboratory values.
Duration of Response (DOR) | Approximately 24 months
  DOR is defined as the time from the date of the first response (CR/PR) until the date of radiological progressive disease or death due to any cause (whichever occurs first).
Progression Free Survival(PFS) | Approximately 24 months
  PFS is defined as the duration from the subject's first dose of the investigational product to the first imaging confirmation of radiological progressive disease or death due to any cause (whichever occurs first).
Overall Survival (OS) | Approximately 24 months
  OS is defined as the duration from the first dose of the investigational product to the time point when death occurs due to any cause.
Maximum concentration (Cmax) | Approximately 24 months
  Cmax will be derived from the PK serum samples collected.
Time of the maximum concentration (Tmax) | Approximately 24 months
  Tmax will be derived from the PK serum samples collected.
Terminal elimination half-life (T1/2) | Approximately 24 months
  T1/2 will be derived from the PK serum samples collected.
Clearance (CL) | Approximately 24 months
  CL will be derived from the PK serum samples collected.
Apparent volume of distribution during the terminal phase (Vz) | Approximately 24 months
  Vz will be derived from the PK serum samples collected.
Number of anti-drug antibody (ADA) Positive Participants | Approximately 24 months
  Immunogenicity will be measured by the number of participants that are ADA positive.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China